CLINICAL TRIAL: NCT02426736
Title: Effect of Dexamethasone Dose and Route on Duration of Interscalene Brachial Plexus Block for Outpatient Arthroscopic Shoulder Surgery - A Randomized Controlled Trial
Brief Title: Effect of Dexamethasone Dose and Route on Duration of Interscalene Block After Outpatient Shoulder Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Thomas Mutter, Assistant Professor of Anesthesia, University of Manitoba
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B2015:016
Record Dates: First submitted 2015-04-14; First posted 2015-04-27 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2017-10

CONDITIONS: Pain, Postoperative; Disorder of Shoulder
Keywords: Shoulder Joint; Arthroscopy; Ambulatory surgical procedures; Pain, Postoperative; Brachial Plexus Block; Corticosteroid; Dexamethasone; Bupivacaine; Perineural
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Low dose intravenous dexamethasone (Active Comparator): 4 milligrams dexamethasone administered once intravenously with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Procedure: Interscalene brachial plexus block
- High dose intravenous dexamethasone (Active Comparator): 8 milligrams dexamethasone administered once intravenously with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Procedure: Interscalene brachial plexus block
- Low dose perineurial dexamethasone (Active Comparator): 4 milligrams dexamethasone administered once perineurally with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Procedure: Interscalene brachial plexus block
- High dose perineurial dexamethasone (Active Comparator): 8 milligrams dexamethasone administered once perineurally with a 30 millilitres 0.5% bupivacaine interscalene brachial plexus block
  Interventions: Drug: Dexamethasone; Drug: Bupivacaine; Procedure: Interscalene brachial plexus block

INTERVENTIONS:
Drug: Dexamethasone
Drug: Bupivacaine
Procedure: Interscalene brachial plexus block — Performed with real time ultrasound guidance.

SUMMARY:
In this factorial design study, 280 participants having outpatient, arthroscopic shoulder surgery will be randomized into 4 equal sized groups. All participants will receive a standardized interscalene brachial plexus block and 4mg or 8mg of dexamethasone given by the intravenous or perineural (by the nerve with the nerve block) route just prior to their surgery. The purpose of this study is to determine which dose and route of dexamethasone provides the longest duration of pain control and the fewest side effects after surgery. The investigators hypothesize that giving dexamethasone by the perineural route, and by higher doses, will result in the longer durations of pain control, without increased side effects.

DETAILED DESCRIPTION:
BACKGROUND & RATIONALE Interscalene brachial plexus blockade (ISB) has emerged as the choice method of analgesia for arthroscopic shoulder surgery performed on an outpatient basis. The ISB is typically administered as a single injection of local anesthetic prior to surgery. Benefits include reduced pain, opioid consumption and postoperative nausea and vomiting on the first postoperative day. However, the limited duration of analgesia with a single injection of local anesthetic, typically 12 to15 hours, is inadequate for many patients. Recent interest in prolonging the analgesic duration of single injection ISB has been focused on the addition of various adjuncts to the local anesthetic, with varying degrees of success.

Dexamethasone is the most promising of these adjuncts, with both perineural and intravenous administration consistently resulting in increased analgesic duration, by as much as two-fold. Nevertheless, it would seem prudent to administer perineural adjuncts at the lowest effective dose and only if they offer significant benefit over other routes of administration.

The multiple small clinical studies published to date have used dexamethasone doses between 4 and 10mg for both intravenous and perineural routes. Attributing differences in results between any of these studies to the dose and route of dexamethasone administered is not possible due to differences in drugs, doses, study populations and methodology. Most importantly, no study has compared two different doses of dexamethasone and the only two studies that compared the intravenous and perineural routes arrived at different conclusions. Thus, the effect of dexamethasone dose and route on the analgesic duration of interscalene block remains unclear, with multiple recent editorials and meta-analyses calling for further study. In light of these gaps in the evidence, a trial elucidating the effect of dose and route of administration of dexamethasone on analgesic duration of ISB is required. This is the focus of our proposed study.

OBJECTIVES AND HYPOTHESES In this factorial design study of outpatients undergoing elective arthroscopic shoulder surgery with interscalene brachial plexus block (ISB), the investigators will compare perineural and intravenous administration of dexamethasone at high (8mg) and low (4mg) doses. The investigators hypothesize that high doses and the perineural route will provide significantly longer duration of analgesia, without significant statistical interaction between dose and route of administration.

METHODS This single-centre, factorial design, double-blinded, randomized controlled superiority trial has four parallel groups and 1:1:1:1 randomization. Consenting and eligible adult ambulatory patients undergoing arthroscopic shoulder surgery will receive preoperative, ultrasound guided ISB with 30 millilitres (mL) of 0.5% bupivacaine and 4mg or 8mg of preservative free dexamethasone either intravenous or perineural. The remainder of the intraoperative and postoperative care is at the discretion of the attending anesthesiologist and surgeon. Based on previous work, with 70 patients per group, the study is at least 90% powered to detect a 3 hour difference in analgesia for dose or route, and a 4 hour synergistic interaction, even with a 5% attrition rate. Outcomes will be assessed by chart review and telephone follow up on postoperative day one, postoperative day 2 (if necessary), and postoperative day 14.

An interim analysis of group standard deviations only will occur after 100 patients have completed the study to determine if the original power calculations were accurate, and if testing for the interaction effect is feasible within the planned sample size of 280 participants. If testing for the interaction of dose and route is not feasible, a new study sample size will be determined, based on the number of participants needed to have 90% power to test the two main effects.

The primary outcome analysis will analyze by intention to treat only those patients who were randomized and did receive an attempt at an interscalene block. A secondary analysis will exclude patients who had a "failed" inter scalene block in the post anesthesia care unit. A tertiary analysis will be a multivariable analysis adjusted for demographics, preoperative naproxen use, use of general anesthesia, cumulative analgesic use and failed inter scalene block.

ELIGIBILITY:
Inclusion Criteria:

* Elective ambulatory surgery patients undergoing arthroscopic shoulder surgery
* Including rotator cuff repair
* Stabilization procedures
* Acromioplasty
* Debridement and distal clavicle excision

Exclusion Criteria:

* Patient refusal, diabetes
* Pregnancy
* Coagulopathy significant enough to be a contraindication to regional anesthesia as determined by the attending anesthesiologist
* Sensitivity to local anesthetics or dexamethasone
* Severe chronic obstructive pulmonary disease
* Contralateral vocal cord paralysis
* Contralateral diaphragmatic paralysis
* Surgical limb brachial plexus neuropathy
* Interscalene block site infection
* Systemic glucocorticoids in the last 2 weeks
* Epidural or intraarticular steroid injection in the past 3 months
* Chronic opioid use defined as daily use for the last two weeks
* International normalized ratio (INR) > 1.5
* Active peptic ulcer disease
* End-stage renal disease
* Cirrhotic liver disease
* Previous participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2015-06-25 (Actual); Primary Completion 2016-07-12 (Actual); Study Completion 2017-01-12 (Actual)

PRIMARY OUTCOMES:
Duration of analgesia after interscalene block | Time-to-event outcome measure, assessed up to the end of postoperative day 2 (approximately 60 hours from performance of the block).
  Time from block performance to the first time shoulder pain was experienced after the surgery, rounded to the nearest 0.1 hours, as reported by the participant at telephone follow-up on postoperative day one, or if necessary, postoperative day 2.

SECONDARY OUTCOMES:
Block Success or Failure | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after the performance of the block.
  The block will be considered "failed" if the patient required opioid analgesia for surgical site pain during their stay in the post anesthesia care unit, as determined by the patient's nurse. At our facility, patients are discharged home directly from the post anesthesia care unit.
Severity of pain at the time the primary outcome occurred, measured on an 11-point numerical rating score. | Assessed at the time that the primary outcome occurs, an expected average of 20 hours after performance of the block.
  11-point numerical rating score, with integers from 0 to 10 where 0 represents no pain and 10 represents worst imaginable pain. As reported by telephone follow up.
Cumulative Analgesic Consumption in the post anesthesia care unit, measured as equivalent milligrams of morphine. | "Change" outcome measure: From admission to the post anesthesia care unit (an expected average of 3 hours after performance of the block), to discharge from the post anesthesia care unit (an expected average of 5 hours after performance of the block).
Cumulative Analgesic Consumption from post anesthesia care unit discharge until the time the primary outcome occurred, measured as equivalent milligrams of morphine. | "Change" outcome measure: From discharge from the post anesthesia care unit (an expected average of 5 hours after performance of the block), to the occurrence of the primary outcome (an expected average of 20 hours after performance of the block).
Postoperative Nausea and/or vomiting measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one.
  11-point numerical rating score, with integers from 0 to 10 where 0 represents the symptom was completely absent and 10 represents the symptom was present the entire time since arrival to the post anesthesia care unit.
First postoperative night Sleep Quality, measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one.
  11-point numerical rating score, with integers from 0 to 10 where 0 represents a very poor sleep and 10 represents a very restful night's sleep.
Observed postoperative Dyspnea, as recorded in the post anesthesia care unit record. | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after performance of the block.
  As observed and recorded by the post anesthesia care unit nurse during the patient's stay in the post anaesthesia care unit.
Subjective postoperative Dyspnea, measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one.
  11-point numerical rating score, with integers from 0 to 10 where 0 represents the symptom was completely absent and 10 represents the symptom was present the entire time since admission to the post anesthesia care unit.
Restlessness and/or Anxiety, measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one.
  11-point numerical rating score, with integers from 0 to 10 where 0 represents the symptom was completely absent and 10 represents the symptom was present the entire time since admission to the post anesthesia care unit.
Motor and/or Sensory Block Dissatisfaction, measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one
  11-point numerical rating score, with integers from 0 to 10 where 10 represents complete dissatisfaction and 0 represents no dissatisfaction.
Likelihood of choosing this method of analgesia again, measured on an 11-point numerical rating score. | Assessed at telephone follow up on postoperative day one
  11-point numerical rating score, with integers from 0 to 10 where 10 "would for sure choose this method again", and 0 represents "would for sure not choose this method again".
Unplanned Postoperative Hospital Admission, as reported at telephone follow up or chart review. | Assessed at telephone follow up and chart review on postoperative day one.
  Transfer or admission to hospital during the postoperative period between admission to the post anesthesia care unit and telephone follow up on postoperative day one.
New Persistent Neurologic Symptoms | Assessed at postoperative day 14.
  Patient will be asked whether they are experiencing any tingling, numbness or weakness in the surgical limb, or hoarseness or dyspnea. Patients answering yes to any of the above will be reassessed at 6 months postoperatively.
Post anesthesia care unit length of stay in minutes | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after performance of the block.
  Amount of time between admission and discharge from the post anesthesia care unit.

OTHER OUTCOMES:
Intraoperative and post anesthesia care unit use of cardiovascular medications, as recorded in the patient's chart. | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after the performance of the block.
  The use of Intraoperative vasopressors, inotropes, antimuscarinics or antihypertensives at any time between the performance of the block and discharge from the post anesthesia care unit.
Adverse events previously related to the inter scalene block and unlikely related to dexamethasone, as recorded in the patient's chart. | Assessed at discharge from the post anesthesia care unit, an expected average of 5 hours after the performance of the block.
  The occurrence of seizure, systemic local anesthetic toxicity, pneumothorax, hemothorax, epidural spread of local anesthetic, or hoarse voice at any time between the performance of the block and discharge from the post anesthesia care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Mutter, MD MSc, Principal Investigator — Assistant Professor
Locations (1):
- Pan Am Surgical Centre, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Fortier J, Chung F, Su J. Unanticipated admission after ambulatory surgery--a prospective study. Can J Anaesth. 1998 Jul;45(7):612-9. doi: 10.1007/BF03012088. PMID 9717590
- [Background] Hughes MS, Matava MJ, Wright RW, Brophy RH, Smith MV. Interscalene brachial plexus block for arthroscopic shoulder surgery: a systematic review. J Bone Joint Surg Am. 2013 Jul 17;95(14):1318-24. doi: 10.2106/JBJS.L.01116. No abstract available. PMID 23864181
- [Background] Fredrickson MJ, Krishnan S, Chen CY. Postoperative analgesia for shoulder surgery: a critical appraisal and review of current techniques. Anaesthesia. 2010 Jun;65(6):608-624. doi: 10.1111/j.1365-2044.2009.06231.x. PMID 20565394
- [Background] Wu CL, Rouse LM, Chen JM, Miller RJ. Comparison of postoperative pain in patients receiving interscalene block or general anesthesia for shoulder surgery. Orthopedics. 2002 Jan;25(1):45-8. doi: 10.3928/0147-7447-20020101-15. PMID 11811241
- [Background] Boezaart AP. Continuous interscalene block for ambulatory shoulder surgery. Best Pract Res Clin Anaesthesiol. 2002 Jun;16(2):295-310. doi: 10.1053/bean.2002.0239. PMID 12491559
- [Background] Choi S, Rodseth R, McCartney CJ. Effects of dexamethasone as a local anaesthetic adjuvant for brachial plexus block: a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2014 Mar;112(3):427-39. doi: 10.1093/bja/aet417. Epub 2014 Jan 10. PMID 24413428
- [Background] Bailard NS, Ortiz J, Flores RA. Additives to local anesthetics for peripheral nerve blocks: Evidence, limitations, and recommendations. Am J Health Syst Pharm. 2014 Mar 1;71(5):373-85. doi: 10.2146/ajhp130336. PMID 24534592
- [Background] Brummett CM, Williams BA. Additives to local anesthetics for peripheral nerve blockade. Int Anesthesiol Clin. 2011 Fall;49(4):104-16. doi: 10.1097/AIA.0b013e31820e4a49. PMID 21956081
- [Background] Vieira PA, Pulai I, Tsao GC, Manikantan P, Keller B, Connelly NR. Dexamethasone with bupivacaine increases duration of analgesia in ultrasound-guided interscalene brachial plexus blockade. Eur J Anaesthesiol. 2010 Mar;27(3):285-8. doi: 10.1097/EJA.0b013e3283350c38. PMID 20009936
- [Background] Cummings KC 3rd, Napierkowski DE, Parra-Sanchez I, Kurz A, Dalton JE, Brems JJ, Sessler DI. Effect of dexamethasone on the duration of interscalene nerve blocks with ropivacaine or bupivacaine. Br J Anaesth. 2011 Sep;107(3):446-53. doi: 10.1093/bja/aer159. Epub 2011 Jun 14. PMID 21676892
- [Background] Tandoc MN, Fan L, Kolesnikov S, Kruglov A, Nader ND. Adjuvant dexamethasone with bupivacaine prolongs the duration of interscalene block: a prospective randomized trial. J Anesth. 2011 Oct;25(5):704-9. doi: 10.1007/s00540-011-1180-x. Epub 2011 Jun 17. PMID 21681533
- [Background] Kim YJ, Lee GY, Kim DY, Kim CH, Baik HJ, Heo S. Dexamathasone added to levobupivacaine improves postoperative analgesia in ultrasound guided interscalene brachial plexus blockade for arthroscopic shoulder surgery. Korean J Anesthesiol. 2012 Feb;62(2):130-4. doi: 10.4097/kjae.2012.62.2.130. Epub 2012 Feb 20. PMID 22379567
- [Background] Desmet M, Braems H, Reynvoet M, Plasschaert S, Van Cauwelaert J, Pottel H, Carlier S, Missant C, Van de Velde M. I.V. and perineural dexamethasone are equivalent in increasing the analgesic duration of a single-shot interscalene block with ropivacaine for shoulder surgery: a prospective, randomized, placebo-controlled study. Br J Anaesth. 2013 Sep;111(3):445-52. doi: 10.1093/bja/aet109. Epub 2013 Apr 15. PMID 23587875
- [Background] Kawanishi R, Yamamoto K, Tobetto Y, Nomura K, Kato M, Go R, Tsutsumi YM, Tanaka K, Takeda Y. Perineural but not systemic low-dose dexamethasone prolongs the duration of interscalene block with ropivacaine: a prospective randomized trial. Local Reg Anesth. 2014 Apr 5;7:5-9. doi: 10.2147/LRA.S59158. eCollection 2014. PMID 24817819
- [Background] De Oliveira GS Jr, Almeida MD, Benzon HT, McCarthy RJ. Perioperative single dose systemic dexamethasone for postoperative pain: a meta-analysis of randomized controlled trials. Anesthesiology. 2011 Sep;115(3):575-88. doi: 10.1097/ALN.0b013e31822a24c2. PMID 21799397
- [Background] Price C, Arden N, Coglan L, Rogers P. Cost-effectiveness and safety of epidural steroids in the management of sciatica. Health Technol Assess. 2005 Aug;9(33):1-58, iii. doi: 10.3310/hta9330. PMID 16095548
- [Background] Latham JM, Fraser RD, Moore RJ, Blumbergs PC, Bogduk N. The pathologic effects of intrathecal betamethasone. Spine (Phila Pa 1976). 1997 Jul 15;22(14):1558-62. doi: 10.1097/00007632-199707150-00004. PMID 9253088
- [Background] Williams BA, Hough KA, Tsui BY, Ibinson JW, Gold MS, Gebhart GF. Neurotoxicity of adjuvants used in perineural anesthesia and analgesia in comparison with ropivacaine. Reg Anesth Pain Med. 2011 May-Jun;36(3):225-30. doi: 10.1097/AAP.0b013e3182176f70. PMID 21519308
- [Background] Sondekoppam RV, Uppal V, Ganapathy S. Intravenous or perineural dexamethasone for interscalene brachial plexus block: the equivalence not yet proven. Br J Anaesth. 2014 Jan;112(1):175-6. doi: 10.1093/bja/aet454. No abstract available. PMID 24318708
- [Background] Fields KG, YaDeau J. Dexamethasone for increasing analgesic duration of single-shot inter-scalene block. Br J Anaesth. 2014 Jan;112(1):176-7. doi: 10.1093/bja/aet455. No abstract available. PMID 24318710
- [Background] Martinez V, Fletcher D. Dexamethasone and peripheral nerve blocks: on the nerve or intravenous? Br J Anaesth. 2014 Sep;113(3):338-40. doi: 10.1093/bja/aeu144. Epub 2014 Jun 6. No abstract available. PMID 24907282
- [Background] Albrecht E, Kern C, Kirkham KR. Perineural vs intravenous administration of dexamethasone: more data are available. Br J Anaesth. 2015 Jan;114(1):160. doi: 10.1093/bja/aeu421. No abstract available. PMID 25500397
- [Background] Albrecht E, Kern C, Kirkham KR. A systematic review and meta-analysis of perineural dexamethasone for peripheral nerve blocks. Anaesthesia. 2015 Jan;70(1):71-83. doi: 10.1111/anae.12823. Epub 2014 Aug 14. PMID 25123271
- [Derived] Holland D, Amadeo RJJ, Wolfe S, Girling L, Funk F, Collister M, Czaplinski E, Ferguson C, Leiter J, Old J, MacDonald P, Dufault B, Mutter TC. Effect of dexamethasone dose and route on the duration of interscalene brachial plexus block for outpatient arthroscopic shoulder surgery: a randomized controlled trial. Can J Anaesth. 2018 Jan;65(1):34-45. doi: 10.1007/s12630-017-0989-7. Epub 2017 Nov 10. PMID 29127558